CLINICAL TRIAL: NCT05923255
Title: Laparoscopic Ileocecal-Sparing Right Hemicolectomy for Cancer of the Hepatic Flexure and Proximal Transverse Colon -- A Prospective, Multicenter Randomized Control Clinical Trial
Brief Title: LISH Trial for the Hepatic Flexure and Proximal Transverse Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCCZ-S03
Record Dates: First submitted 2023-05-30; First posted 2023-06-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Flexure Colon Cancer; Proximal Transverse Colon Cancer
Keywords: hepatic flexure colon cancer; proximal transverse colon cancer; ileocecus-sparing; laparoscopic right hemicolectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LISH （Laparoscopic Ileocecal-Sparing Right Hemicolectomy）group (Experimental): In LISH group, patients suffering from cancer of the hepatic flexure and proximal transverse colon will be undergoing a novel radical right hemicolectomy technique that allows for the preservation of the ileocecal region.
  Interventions: Procedure: LISH （Laparoscopic Ileocecal-Sparing Right Hemicolectomy）
- TRH （Traditional Right Hemicolectomy）group (Active Comparator): In TRH group, patients suffering from cancer of the hepatic flexure and proximal transverse colon will be undergoing the traditional radical right hemicolectomy.
  Interventions: Procedure: TRH（Traditional Laparoscopic Right Hemicolectomy）

INTERVENTIONS:
Procedure: LISH （Laparoscopic Ileocecal-Sparing Right Hemicolectomy） — Preserve the ileocolic blood vessels, and perform dissection of lymph node groups 203, 202, and 201d along the root of ICV(Ileocolic artery)/ICA(Ileocolic vein). Group 201d lymph nodes are defined as the distal lymph nodes of the ileocolic vessels (colonic branch). Use an intracavitary cutting and sealing device to transect the proximal colon along the predetermined margin, and transect the transverse colon at 10cm distal to the tumor. Perform ileocecal-transverse colonic anastomosis.
  Arms: LISH （Laparoscopic Ileocecal-Sparing Right Hemicolectomy）group
Procedure: TRH（Traditional Laparoscopic Right Hemicolectomy） — Transect the root of the ileocolic vessels and perform dissection of lymph node groups 203, 202, and 201; sever the roots of the right colic and middle colic vessels, and clear the surrounding lymphoadipose tissue (lymph node groups 211/212/213 and 221/222/223). Transect the transverse colon 10cm distal to the tumor and cut the terminal ileum 10cm from the ileocecal junction. Perform ileum-to-transverse colon anastomosis.
  Arms: TRH （Traditional Right Hemicolectomy）group

SUMMARY:
The goal of this clinical trial is to compare the long-term outcomes of Laparoscopic Ileocecal-Sparing Right Hemicolectomy(LISH) compared to traditional laparoscopic right hemicolectomy(TRH) in the treatment of hepatic flexure colon cancer and proximal transverse colon cancer.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-labeled, randomized controlled clinical trial. The enrolled patients will be randomly assigned to either the LISH or TRH group in a 1:1 ratio and will receive the corresponding surgery. The primary endpoint: 3-year disease free survival. The second endpoint: 30-day perioperative complications, pathological outcomes (specimen quality, positive resection margin rate, number of lymph nodes retrieved, and lymph node positivity rate), histological prognostic indicators (planned for superiority testing: 1-, 3-, and 5-year rates of newly detected polyps and adenomas on colonoscopy), quality of life (planned for superiority testing: Gastrointestinal Symptom Rating Scale [GSRS] score and EQ-5D-5L score), and 5-year overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-75 years old
2. ASA classification ≤III
3. Colon adenocarcinoma confirmed by endoscopy and pathological biopsy
4. Enhanced abdominal CT indicating the primary lesion is located in the hepatic flexure of the colon or proximal transverse colon (proximal 1/3 of the transverse colon)
5. Preoperative clinical staging: TanyNanyM0
6. Patients able to understand the study protocol, willing to participate in the research, and providing written informed consent

Exclusion Criteria:

1. Preoperative examination indicates synchronous multiple primary colorectal cancers or other diseases requiring bowel segment resection
2. Preoperative imaging or intraoperative exploration reveals: 1) tumor involving surrounding organs requiring combined organ resection; 2) presence of distant metastasis; 3) inability to perform R0 resection; 4) fused and fixed lymph nodes at the root of the ileocolic vessels
3. Additional radical surgery following Endoscopic Mucosal Resection (EMR) and Endoscopic Submucosal Dissection (ESD) procedures
4. History of any other malignant tumor within the last 5 years or familial adenomatous polyposis, except for cured in situ cervical cancer, basal cell carcinoma, papillary thyroid carcinoma, or skin squamous cell carcinoma
5. Presence of bowel obstruction, bowel perforation, or intestinal bleeding requiring emergency surgery
6. Patients unsuitable for or unable to tolerate laparoscopic surgery
7. Pregnant or lactating women
8. Patients with a history of psychiatric disorders
9. Patients who have received neoadjuvant therapy prior to surgery
10. Patients deemed unsuitable for the study by MDT discussion
11. Patients unable to understand the study's conditions and objectives, and refusing to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2023-05-14 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2031-05-14 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years
  the time from enrollment until disease relapse or death from any cause 3 years after surgery

SECONDARY OUTCOMES:
Perioperative complications | up to 30 days after surgery
  Complications occurring within 30 days after surgery. Perioperative complications are classified according to the Clavien-Dindo classification system and include intraoperative, short-term, and long-term postoperative complications. The following events are considered serious perioperative complications: hemorrhage requiring transfusion of >4 units of packed red blood cells; postoperative complications necessitating emergent surgical intervention; severe infection (as defined by the American College of Chest Physicians/Society of Critical Care Medicine 1992 criteria); and deaths attributable to the surgical procedure. These should be reported within 30 days postoperatively.
Quality of the specimen | up to 2 weeks after surgery
  The data included specimen quality, positive margin rate, number of harvested lymph nodes and positive lymph nodes
Incidence rates of polyps and adenomas | 5 years
  the incidence rates of polyps and adenomas as seen on colonoscopy at 1, 3 and 5 years after surgery respectively.
Scores of quality of life | 3 years
  measured by scores from the Gastrointestinal Symptom Rating Scale (GSRS) at 1, 2, and 3 years after surgery respectively, and scores from the EQ-5D-5L Quality of Life Scale at 1, 2, and 3 years after surgery respectively.
Scores from the EQ-5D-5L Quality of Life Scale | 3 years
  scores from the EQ-5D-5L Quality of Life Scale at 1, 2, and 3 years after surgery respectively.
5-year overall survival rate (OS) | 5 years
  The proportion of patients who survived 5 years after surgery, taking into account any cause of death.

OTHER OUTCOMES:
Conversion Rate from Laparoscopic to Open Surgery | Intraoperative period
  The proportion of laparoscopic surgeries that are converted to open surgeries due to intraoperative complications, technical challenges, or other clinical reasons.
LISH Surgery Completion Rate | Intraoperative period
  The proportion of patients in whom the LISH procedure is successfully completed without conversion to TRH or other alternative surgical approaches.
Minimal Residual Disease (MRD) via Circulating Tumor DNA (ctDNA) | Preoperative (7 days), postoperative (7 days), and 3 months post-surgery
  Detection of MRD using circulating tumor DNA (ctDNA) as a biomarker.
Short- and Long-Term Changes in Gut Microecology | Preoperative, postoperative 3 months, 6 months and 12 months
  Analysis of gut microbiota, epithelial cells, stromal cells, immune cells, and metabolic products using fecal samples and intestinal biopsy tissues.
Glycemic Metabolic Indicators - Hemoglobin A1c (HbA1c) | Preoperative, 3 months, 6 months, and 12 months post-surgery
  Measurement of glycated hemoglobin (HbA1c) levels to assess long-term glycemic control.
Oral Glucose Tolerance Test (OGTT) | Preoperative, 3 months, 6 months, and 12 months post-surgery
  Evaluation of glucose metabolism by measuring blood glucose and insulin levels at 0, 30, 60, 120 minutes after oral glucose administration.
Insulin Resistance (HOMA-IR) | Preoperative, 3 months, 6 months, and 12 months post-surgery
  Calculation of insulin sensitivity using fasting glucose and insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (29):
- China (29):
  - the First Affiliated Hospital of Bengbu Medical Collage, Bengbu, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Academy of medicine Scenice, Beijing, Beijing Municipality
  - the First Affiliated Hospital of Chongqing Medical Collage, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Hospital Medical Union University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technolog, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Jiangsu province hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated of The Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality
  - The first affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi
  - West China Hospital of Sichuang University, Chengdu, Sichuan
  - The Cancer Hospital Affiliated of The Xingjiang University Medical School, Xinjiang, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Second Affiliated Hospital Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of medicien, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No